CLINICAL TRIAL: NCT00208559
Title: Ziprasidone in Children With Autism: A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Richard P. Malone, Drexel University College of Medicine
Organization: Drexel University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00936
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Autism
Keywords: Autism; Pervasive Developmental Disorder; Ziprasidone; Adolescents
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 Open Label (Other): Open Label
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — Ziprasidone 40mg to 60mg per day, individually titrated
  Other Names: Geodon

SUMMARY:
The purpose of this study is to see if the drug, ziprasidone, is effective in treating problems in adolescent associated with autism.

DETAILED DESCRIPTION:
I. SPECIFIC AIMS

1. To investigate the safety of clinical use of ziprasidone in children
2. To investigate the dosages that have been employed clinically.

II. BACKGROUND AND SIGNIFICANCE

Ziprasidone, a recently released atypical agent is likely to be as effective as other neuroleptics in treating psychiatric symptoms in children, but may have the considerable health advantage of not causing weight gain. Ziprasidone administration has been associated with prolongation of the QTc interval (mean=20 msec), an electrocardiographic measure of ventricular repolarization (Federal Drug Administration, 2000). There are no reports regarding the use of ziprasidone in autism, and data regarding the safety and efficacy of ziprasidone in children is extremely limited. The only published study of ziprasidone in children found that it was safe and effective in treating Tourette's syndrome in children aged 7 to 17 years of age (Sallee et al, 2000). Because children are being treated with ziprasidone despite a paucity of safety data, it is important to begin to collect and review available data, including that from clinical usage. Some children who receive services within the Child and Adolescent Psychiatric Services of Drexel University College of Medicine have been treated with ziprasidone. The charts of the children and adolescents will contain data regarding exposure to ziprasidone and laboratory data and ECG's that can be reviewed to determine whether ziprasidone treatment has been associated with changes in weight, laboratory values and ECG's. We propose to review the charts of patients who have been treated with our services since March 1, 2001 XXX because such patients may have been exposed to ziprasidone (ziprasidone received FDA approval on February 5, 2001).

III. DESIGN AND METHODS

A. Setting: The setting for this study will be the Specialty Clinic for Pervasive Developmental Disorders, part of the Child and Adolescent Psychiatry Outpatient Clinic at Eastern Pennsylvania Psychiatric Institute.

B. Subjects: Subjects will be 15 children and adolescents who meet the DSM-IV Criteria for Pervasive Developmental Disorder.

C. Design: This is a 6-week pilot study employing open treatment with ziprasidone. Subjects will be rated at baseline and thereafter assessed weekly.

D. Medication: Subjects will be treated openly with ziprasidone. Should untoward effects occur, the dosage of the medication will be reduced or the medication will be discontinued, as clinically appropriate. Subjects will not receive other concomitant psychotropic medication during the study. Medication will be taken concomitant with food.

Ziprasidone Dosing Strategy: Ziprasidone tablets (5, 10, and 20 mg) will be employed for the study. The dosage range for ziprasidone will be 5 mg/day to 40 mg/day. Every effort will be made to reach and maintain a therapeutic dosage by week four of the treatment phase.

1. For subjects who weigh less than 25 kg, starting dosage will be 5 mg/every other day. After 3 days, the dosage can be increased to 5 mg. By week 2, subjects can be increased to 20 mg/day. Thereafter, dosage increases can be made in up to 20 mg increments weekly.
2. For subjects who weigh greater than 25 kg, the starting dosage will be 5 mg/day. After three days, the dosage can be increased to 10 mg/day. By week two, subjects can be increased to 20 mg/day. Thereafter, dosage increases can be made in up to 20 mg increments weekly as needed.

Note: Should 5 mg tablets not be available, the dosing schedule will be altered to have a starting dosage of 10 mg, and dosage increases will be made in 10 mg increments.

F. Measures

1. Primary efficacy measure: The Clinical Global Impressions (CGI; Psychopharmacology Bulletin, 1985). The efficacy of treatments can be judged on their ability to enhance global functioning, an assessment that is particularly relative in a pilot study. The CGI consists of three global scales measuring severity of illness, global improvement, and drug effect, and has been useful in measuring drug treatment effect in this population (see Campbell and Palij, 1985). The PI and another trained rater will complete this scale. Although only members of the research team generally complete this scale, it will additionally be completed by the subject's parent/caretaker. Having it completed by the parent/caretaker will take only minutes and may result in useful data. This measure will be completed weekly beginning at baseline.
2. Secondary efficacy measure: Children's Psychiatric Rating Scale (Psychopharmacology Bulletin, 1985). The CPRS was developed by the Psychopharmacology Branch of the NIMH to rate childhood psychopathology. Each of the items is rated from "1" (not present) to "7" (extremely severe). The first 28 items of this scale require no verbal response on the part of the subject, making them appropriate for rating children and adolescents with Pervasive Developmental Disorder. Of these 28 items, 14 are particularly relevant in autism (see Campbell and Palij, 1985): they assess the symptoms for which drug treatment is indicated including hyperactivity, aggression, self-abusive behavior, temper tantrums, lability of mood, irritability, social withdrawal, and stereotypies. A composite sum of these 14 items, the CPRS-14, will be constructed and employed as a secondary outcome measure, a procedure used by a number of investigators (Anderson et al, 1989; Campbell et al, 1986, 1989, 1993; Findling et al, 1997; Sanchez et al, 1996). We analyzed our data using the CPRS-14; the ICC was 0.8978. In addition, 4 factors derived from these 14 items will be examined. They include: autism, anger/uncooperativeness, hyperactivity, and speech deviance (Overall and Campbell, 1988). This measure will be completed at baseline and at the end of treatment.
3. Safety measures: (1) A physical exam will be completed at baseline. (2) Height, weight, blood pressure, and pulse will be obtained and recorded at baseline and at each visit during the study. (3) The following laboratory measures will be obtained at baseline and repeated at the end of the treatment phase: complete blood count with differential, liver functions, and electrocardiogram. Serum prolactin will be obtained at baseline and at the end of the treatment phase. These laboratory studies will be repeated at the end of the treatment phase of the study. Any other clinically appropriate tests and evaluations will also be completed whenever needed.

Untoward effects will be measured and recorded at each visit employing the following measures: (1) Dosage Record and Treatment Emergent Symptom Scale (DOTES); (2) Treatment Emergent Symptoms Scale (TESS); (3) Abnormal Involuntary Movement Scale (AIMS) (all from Psychopharmacology Bulletin, 1985); and (4) the Neurologic Rating Scale (Simpson and Angus, 1970). The DOTES and TESS measure a wide range of possible untoward effects. The AIMS measures dyskinesias. The Neurologic Rating Scale measures other forms of extrapyramidal effects that can occur with neuroleptics such as dystonias, parkinsonian effects, and akathisia.

G. Procedures: All patients appropriate to the study and their parent/caretakers will be approached and informed consent and assent (in subjects under 14 years) will be obtained. Subjects meeting the Inclusion Criteria, but not the Exclusion Criteria, will enter the baseline period of the study.

Baseline (week 0): Subjects will be rated at baseline employing the CGI and the CPRS.

End of Treatment (week 6): At the end of the treatment period, subjects will again be rated employing the CGI and the CPRS (selected items).

In addition, each subject will be rated on the CGI at each visit so that data from the last visit is available should the subject terminate the study prematurely. If it is known that a subject will terminate the study at a visit before week 6, the subject will be rated with the CGI and the CPRS at that visit.

All safety measures will be completed at each visit. Laboratory measures and EKG will be obtained in the morning.

I. Analysis: This is a pilot study whose purpose is to get initial safety and efficacy data with ziprasidone in children with autism. We will perform an ANOVA, repeated measures, for CGI severity scores, the CPRS-14 and the CPRS factors. Similar analyses will be performed for safety measures including for weight, prolactin and other laboratory measures, and EKG indices.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism (DSM-IV) made by a boarded child and adolescent psychiatrist.
* Males and females.
* Aged 12 to 18 years.
* Clinical judgment that medication treatment for autism is indicated.

Exclusion Criteria:

* Major medical problems including cardiac, liver, endocrine, or renal diseases.
* History of seizure disorder or gross neurological deficit.
* Baseline QTC greater than 425 msec.
* Concomitant treatment with psychotropic medication.
* History of prior exposure to ziprasidone.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2002-02; Primary Completion 2005-06 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions | Week 6

SECONDARY OUTCOMES:
Children's Psychiatric Rating Scale | Baseline, Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Malone, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Drexel University College of Medicine at Friends Hospital, Philadelphia, Pennsylvania, United States